CLINICAL TRIAL: NCT00005407
Title: Statistical Analysis of Pediatric Task Force Data Base
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4324; R03HL046212 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To define pediatric sex-specific blood pressure percentiles that were a function of both age and height. Also, to define the precise age at which blood pressure distributions for different racial groups diverged.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension is a well-recognized risk factor for cardiovascular disease in adults. Furthermore, many studies have shown that there is tracking among longitudinal pediatric blood pressure determinations. An important unresolved goal in pediatric hypertension research is to define at what level of pediatric blood pressure is a child at increased risk for adult hypertension. When the grant was awarded in February 1991, there had been two NHLBI Task Forces in Blood Pressure Control in Children which had published reports in 1977 and 1987. One of the goals of each task force was to define appropriate percentiles for blood pressure in children. In the Second Task Force Report, results from nine large epidemiologic studies were combined into a data base with more than 70,000 readings from which blood pressure percentiles were derived as a function of age and sex. However, many research workers stated that height is more strongly related to blood pressure than age and have urged that Normative data for pediatric blood pressure be demarcated by height rather than age.

DESIGN NARRATIVE:

Blood pressure percentiles were constructed that were a function of age, sex, race, and height, thus providing a more comprehensive profile of pediatric blood pressure distributions than any previously published work.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-02; Study Completion 1993-01 (Actual)